CLINICAL TRIAL: NCT05645224
Title: Pilot Feasibility Clinical Trial of Virtual Reality for Pain Management During Repeated Pediatric Laser Procedures
Brief Title: VR-PAT for Pain and Anxiety Management During Pediatric Dermatologic Laser Procedures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Henry Xiang, Professor of Medicine and Center Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00002880
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-03

CONDITIONS: Procedural Anxiety; Procedural Pain
Keywords: Laser; Dermatology; Virtual Reality; VR
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention group (VR-PAT) or the control group (same VR google without game) at the first laser procedure and will then cross-over to the alternative group for the second laser procedure.
Who Masked: Investigator
Masking Description: Researcher conducting the post-procedural survey is blinded to the group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-PAT (Experimental): Participant wears the Pico Neo 3 Pro Eye headset and actively plays the VR-PAT game.
  Interventions: Other: VR-PAT
- Control (No Intervention): Participant wears the Pico Neo 3 Pro Eye headset to protect eyes, but it is not turned on.

INTERVENTIONS:
Other: VR-PAT — Virtual Reality Pain Alleviation Therapy (VR-PAT) played on a Pico Neo 3 Pro Eye device
  Arms: VR-PAT

SUMMARY:
This study will assess the feasibility and efficacy of our Virtual Reality Pain Alleviation Therapy (VR-PAT) for pain management during pediatric and young adult outpatient laser procedures and evaluate the impact of VR use on reducing anxiety in patients undergoing dermatologic laser procedures. The investigators hypothesize that patients using VR-PAT will report less pain and anxiety during the laser procedure than patients who do not play the game.

DETAILED DESCRIPTION:
In this two-group crossover randomized clinical trial, patients will be randomly assigned to either the VR-PAT intervention group or control group (same VR google without game) at the first laser procedure and will then cross-over to the alternative group for the second laser procedure. Survey questions to assess pain and anxiety and control for confounding factors will be asked before and after each procedure.

ELIGIBILITY:
Inclusion Criteria:

* dermatology patients (5+ years) who are undergoing first laser procedure at the Nationwide Children's Outpatient Laser
* have a legal guardian present for patients less than 18 years old for the procedure (for informed consent)
* can communicate orally

Exclusion Criteria:

* any wounds that may interfere with study procedures
* usage of a diode laser (VR safety has not been established yet)
* vision, hearing, or cognitive/motor impairments preventing valid administration of study measures
* history of motion sickness, seizure disorder, dizziness, or migraine headaches precipitated by visual auras
* minors in foster care
* unable to communicate in English
* pregnant women
* prisoners

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in procedural pain | Assessed immediately following each laser procedure
  0-10 Numerical Rating Scale (NRS) (self-reported and caregiver-reported (if <18 years)), 0(min)-10(max), with higher score indicating worse pain. Asked for worst pain, average pain, and time spent thinking about pain.
Change in procedural anxiety | Assessed at 3 time points (prior to entering procedure room, prior to the procedure, and immediately following the procedure) for each laser procedure
  Modified Yale Preoperative Anxiety Scale (mYPAS) (observed by researcher), 23.33(min)-100(max), with higher scores denoting higher levels of anxiety.

SECONDARY OUTCOMES:
Self-reported VR experience | Immediately following laser procedure in VR-PAT group
  0-10 Numerical Rating Scale (NRS) (self-reported - VR-PAT arm only), 0(min)-10(max), with higher score meaning better outcome. Asked for degree of realism, pleasure, and satisfaction with VR.
Nurse-reported utility | Immediately following laser procedure in VR-PAT group
  Binary (Yes/No) questions of whether the nurse found VR-PAT to be helpful and easy to use during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiang, MD, MPH, PhD, MBA, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No